CLINICAL TRIAL: NCT06550843
Title: Mesentery Abnormality to Identify Microscopic Clean Resection and Reduce Postoperative Endoscopic Recurrence in Ileocolic Crohn's Disease
Brief Title: Mesentery Guide Identify Microscopic Clean Resection and Reduces Crohn's Endoscopic Recurrence
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jia Ke, Ph.D, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: Sixth Affiliated Hospital 001
Record Dates: First submitted 2024-08-08; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Crohn Disease; Recurrence
Keywords: Mesentery Guide; Microscopic Clean Resection; Endoscopic Recurrence
MeSH Terms: conditions — Crohn Disease; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- conventional group: In the conventional group, the cutting line was approximately 2cm proximal to the macroscopic lesion where the mucosa and intestinal wall appeared macroscopically normal, regardless of the adjacent mesentery.
- mesentery-guided group (Mes-G): In the Mes-G group, all surgeries were performed by one surgeon team (J.K.) from January 2013 using the following strategy for the proximal division site: the diseased bowel and para-intestinal mesentery were carefully compared by palpation and translucent observation through a shadowless lamp. The comparison was conducted from the diseased bowel towards the normal-appearing region upstream, to identify a point where the hypertrophied mesentery transitioned into normal thickness and softness and became translucent as observed through the shadowless lamp.
  Interventions: Procedure: mesentery-guided division

INTERVENTIONS:
Procedure: mesentery-guided division — In the Mes-G group, all surgeries were performed by one surgeon team (J.K.) from January 2013 using the following strategy for the proximal division site: the diseased bowel and para-intestinal mesentery were carefully compared by palpation and translucent observation through a shadowless lamp. The comparison was conducted from the diseased bowel towards the normal-appearing region upstream, to identify a point where the hypertrophied mesentery transitioned into normal thickness and softness and became translucent as observed through the shadowless lamp.
  Groups: mesentery-guided group (Mes-G)

SUMMARY:
Microscopic clean margin is associated with reduced endoscopic recurrence after bowel resection for ileocolic Crohn's disease (CD). We aimed to investigate whether the extent of creeping fat could help indicate microscopic inflammation beyond naked eye assessment of the bowel wall and reduce endoscopic recurrence after ileocolic resection.

DETAILED DESCRIPTION:
Despite proactive prophylactic treatment administered after surgery for Crohn's disease (CD) patients, early postoperative endoscopic recurrence (EPER) still occurs in 50-80% of patients within six months, increasing the risk of long-term clinical and surgical recurrence. Risk factors for EPER have already been identified, including active smoking, disease behavior, younger age, concomitant perianal disease, prior intestinal resections, and microscopic resection margin positivity. Recently, the influence of microscopic inflammation at the resection margin on EPER has been highlighted by various studies and meta-analysis.

From a surgical perspective, it has become common practice to conservatively resect 2cm width from the gross lesion to lower re-operation risks, while the optimal strategy to attain the microscopic clean margin and minimize EPER remain unclear, considering the limited accuracy of frozen-section examinations. More importantly, the diseased mucosa proximal to the ileal lesion can be healed by preoperative optimization, potentially concealing deeper lesions at the muscularis propria and serosal levels from visual assessment during surgery. Therefore, identifying a macroscopic marker that highly correlates with microscopic inflammation is essential to help locate the clean division.

As a hallmark of CD, the hyperplasia of mesenteric adipose tissue (MAT) or "Creeping fat," was found directly triggered by transmural inflammation and bacterial translocation from CD affected lumen11. Correspondingly, creeping fat has been found to correlate with macroscopic mucosal abnormalities observed after opening the bowel12. However, its relationship with microscopic inflammation, as well as its potential role in determining the division position to achieve better EPER outcomes, remains to be clarified.

ELIGIBILITY:
Inclusion Criteria:

* Localized ileocolic CD

Exclusion Criteria:

* Patients with a stoma,residuallesion ,history of bowel resection,or post-operative abdominalinfection were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the pathological study, we prospectively enrolled consecutive CD patients who underwent ileocolic resections between January 2021 and August 2021 at the 6th Hospital of Sun Yat-Sen University (SYSU6H) For the surgical study, we retrospectively enrolled consecutive CD patients that underwent ileocolic resection from January 2013 to July 2020
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Crohn's Endoscopic Recurrence | 12 months

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Hammoudi N, Cazals-Hatem D, Auzolle C, Gardair C, Ngollo M, Bottois H, Nancey S, Pariente B, Buisson A, Treton X, Fumery M, Bezault M, Seksik P, Le Bourhis L; REMIND Study Group Investigators; Flejou JF, Allez M. Association Between Microscopic Lesions at Ileal Resection Margin and Recurrence After Surgery in Patients With Crohn's Disease. Clin Gastroenterol Hepatol. 2020 Jan;18(1):141-149.e2. doi: 10.1016/j.cgh.2019.04.045. Epub 2019 Apr 28. PMID 31042575
- [Background] Tandon P, Malhi G, Abdali D, Pogue E, Marshall JK, de Buck van Overstraeten A, Riddell R, Narula N. Active Margins, Plexitis, and Granulomas Increase Postoperative Crohn's Recurrence: Systematic Review and Meta-analysis. Clin Gastroenterol Hepatol. 2021 Mar;19(3):451-462. doi: 10.1016/j.cgh.2020.08.014. Epub 2020 Aug 12. PMID 32801016
- [Background] Poredska K, Kunovsky L, Marek F, Kala Z, Prochazka V, Dolina J, Zboril V, Kovalcikova P, Pavlik T, Jabandziev P, Pavlovsky Z, Vlazny J, Mitas L. The Influence of Microscopic Inflammation at Resection Margins on Early Postoperative Endoscopic Recurrence After Ileocaecal Resection for Crohn's Disease. J Crohns Colitis. 2020 Mar 13;14(3):361-368. doi: 10.1093/ecco-jcc/jjz153. PMID 31501878
- [Background] Fazio VW, Marchetti F, Church M, Goldblum JR, Lavery C, Hull TL, Milsom JW, Strong SA, Oakley JR, Secic M. Effect of resection margins on the recurrence of Crohn's disease in the small bowel. A randomized controlled trial. Ann Surg. 1996 Oct;224(4):563-71; discussion 571-3. doi: 10.1097/00000658-199610000-00014. PMID 8857860
- [Result] Muller JM, Keller HW, Erasmi H, Pichlmaier H. Total parenteral nutrition as the sole therapy in Crohn's disease--a prospective study. Br J Surg. 1983 Jan;70(1):40-3. doi: 10.1002/bjs.1800700116. PMID 6402050
- [Result] Regueiro M, Velayos F, Greer JB, Bougatsos C, Chou R, Sultan S, Singh S. American Gastroenterological Association Institute Technical Review on the Management of Crohn's Disease After Surgical Resection. Gastroenterology. 2017 Jan;152(1):277-295.e3. doi: 10.1053/j.gastro.2016.10.039. Epub 2016 Nov 10. No abstract available. PMID 27840073
- [Result] Panes J, Rimola J. Perianal fistulizing Crohn's disease: pathogenesis, diagnosis and therapy. Nat Rev Gastroenterol Hepatol. 2017 Nov;14(11):652-664. doi: 10.1038/nrgastro.2017.104. Epub 2017 Aug 9. PMID 28790453